CLINICAL TRIAL: NCT03749668
Title: Dietary Survey During the First Month After Colorectal Surgery Within an Enhanced Recovery Program
Brief Title: Dietary Survey After Colorectal Surgery Within an Enhanced Recovery Program (DIETERP).
Acronym: DIETERP
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Head of the Anesthesiology department, University of Liege
Other Study IDs: 2018-270
Record Dates: First submitted 2018-11-20; First posted 2018-11-21 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Colorectal Surgery; Calorie Deficiency
Keywords: surgery: colorectal; enhanced recovery; caloric intake; protein intake

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non applicable — no intervention in this observational study

SUMMARY:
This observational study will quantify caloric-protein intake in 75 patients undergoing colorectal surgery within an enhanced recovery program at CHU Liège. A dietary survey will be performed preoperatively and repeated postoperatively via telephone calls on Day + 3, Day + 7; Day + 15, and Day + 30, after leaving the hospital. The deficits observed will be correlated with the medical and surgical characteristics of the patients

DETAILED DESCRIPTION:
For several years, we have been applying the concept of Enhanced Recovery Program (ERP) for colorectal surgery at CHU Liége (Belgium). Since October 2015, the University Hospital of Liège has been labelled as reference center for ERP after colorectal surgery by a French-speaking organization GRACE (French-speaking group for Enhanced Recovery after Surgery; www.grace-asso.fr). Despite the benefits for the patient and the economic benefits of such programs, some criticize ERP arguing that patients are asked to return home too early, while they have not recovered a satisfactory autonomy. Few studies have investigated the comfort and quality of home life of patients who have had ERP. We recently conducted a retrospective study to evaluate this quality of life. It turns out that patients report little postoperative pain, a sufficient degree of autonomy at home, and a high general satisfaction score (> 8.5 on a numerical scale of 0 to 10). However dietary and digestive difficulties were described by about one third of the patients questioned. [6] Others have also reported a caloric-protein deficit during the immediate postoperative period after colorectal surgery, up to the 7th day in some of their patients [7].

Aim of the study. The aim of this study is to assess caloric-protein intake up to one month after colorectal surgery within ERP.

General description. This observational study will quantify caloric-protein intake in 75 patients undergoing colorectal surgery according to an ERP at CHU Liège. A dietary survey will be performed preoperatively and repeated postoperatively via telephone calls on Day + 3, Day + 7; Day + 15, and Day + 30, after leaving the hospital. The deficits observed will be correlated with the medical and surgical characteristics of the patients.

ELIGIBILITY:
Inclusion Criteria:

* any patient scheduled for colorectal surgery within an ERP at CHU Liège

Exclusion Criteria:

* unable to answer the survey (cognitive disorders, bad knowledge of the French language)
* closure of loop ileostomy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any patient schedules for colorectal surgery with the ERP at CHU Liège (Belgium). Patients age must be greater than 18 years. There is no maximum limit of age.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-05-08 (Actual)

PRIMARY OUTCOMES:
calorie and protein intakes | one month after hospital discharge
  Using a dietary survey postoperative intake of calories and protein will be assessed in patients scheduled for colorectal surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Brichant, MD, Principal Investigator — CHU Liege, Belgium
Locations (1):
- University Hospital, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No